CLINICAL TRIAL: NCT02634788
Title: A Phase 3, Randomized, Double Blind, Multiple Dose, Parallel Group, Placebo Controlled Study of Buprenorphine Sublingual Spray (0.5 mg TID, 0.25 mg TID, and 0.125 mg TID) for the Treatment of Moderate to Severe Pain
Brief Title: Study of Buprenorphine Sublingual Spray for the Treatment of Moderate to Severe Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS005-15-062
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: Post-Surgical Pain; Bunionectomy
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Buprenorphine 0.5 mg TID (Experimental): Participants received buprenorphine 0.5 mg sublingual (under the tongue) spray three times daily (TID) for two days.
  Interventions: Drug: Buprenorphine
- Buprenorphine 0.25 mg TID (Experimental): Participants received buprenorphine 0.25 mg sublingual spray TID for two days.
  Interventions: Drug: Buprenorphine
- Buprenorphine 0.125 mg TID (Experimental): Participants received buprenorphine 0.125 mg sublingual spray TID for two days.
  Interventions: Drug: Buprenorphine
- Placebo (Placebo Comparator): Participants received placebo-matching buprenorphine sublingual spray TID for two days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine sublingual spray delivered via single 100 μL spray
  Arms: Buprenorphine 0.125 mg TID; Buprenorphine 0.25 mg TID; Buprenorphine 0.5 mg TID
Drug: Placebo — Placebo-matching buprenorphine sublingual spray delivered via single 100 μL spray
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to evaluate analgesic efficacy of Buprenorphine Sublingual (under the tongue) Spray compared with placebo in participants with postoperative pain after bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* History or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni DeCastro, Study Director — INSYS Therapeutics Inc
Locations (4):
- United States (4):
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo-matching buprenorphine sublingual (under the tongue) spray TID for two days.
- Buprenorphine 0.5 mg TID: Participants received buprenorphine 0.5 mg sublingual spray three times daily (TID) for two days.
Period: Overall Study
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Started | 79 | 81 | 80 | 82
Completed | 75 | 71 | 75 | 77
Not Completed | 4 | 10 | 5 | 5
Not completed — Adverse Event | 0 | 8 | 3 | 1
Not completed — Lack of Efficacy | 4 | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who were treated with the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID | Total
Number analyzed (Participants) | 79 | 81 | 80 | 82 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (14.55) | 43.7 (14.17) | 45.6 (11.78) | 48.4 (11.75) | 45.7 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 64 | 64 | 63 | 254
  Male | 16 | 17 | 16 | 19 | 68

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Summed Pain Intensity Difference (SPID) Over 0 to 48 Hours After Time 0 (NRS SPID-48)
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points up to 48 hours after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum(max)=10 at each time point], and negative numbers indicate an increase in pain [minimum(min)=-10 at each time point]. The overall min and max are -10 and 10 times the number of hours specified; SPID-48 range is -480 to 480. The NRS SPID-48 was analyzed using an analysis of covariance (ANCOVA) model, which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Baseline and 0 to 48 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) Population who did not have missing SPID-48 values. Missing SPID-48 data were not imputed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 75 | 72 | 75 | 77
units on a scale | 89.40 (10.109) | 171.33 (10.316) | 125.58 (10.101) | 124.85 (9.944)
Statistical Analysis 1: Comparison: Placebo vs Buprenorphine 0.5 mg TID; Test type: Other; p < 0.0001, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 81.93, 95% CI 2-sided [53.82 to 110.04], Standard Error of Mean 14.283
Statistical Analysis 2: Comparison: Placebo vs Buprenorphine 0.25 mg TID; Test type: Other; p = 0.0108, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 36.18, 95% CI 2-sided [8.43 to 63.93], Standard Error of Mean 14.099
Statistical Analysis 3: Comparison: Placebo vs Buprenorphine 0.125 mg TID; Test type: Other; p = 0.0120, ANCOVA; The analysis included treatment and site as main effects and Baseline pain intensity as the covariate; LS Mean Difference = 35.46, 95% CI 2-sided [7.86 to 63.05], Standard Error of Mean 14.020

2. Secondary Outcome: NRS Mean Pain Intensity Difference (PID) at 4, 8, 24 and 48 Hours After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug administration) and at multiple time points up to 48 hours after Time 0 (time of administration of the first dose of study drug). NRS PID is defined as the difference in pain at each scheduled timepoint relative to Baseline (PID=pain intensity at baseline - pain intensity at time point). A higher value of NRS PID score indicates a higher decrease in pain from Baseline.
Time Frame: Baseline and 4, 8, 24 and 48 hours after Time 0
Population: All randomized participants from the ITT Population with data available at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
units on a scale
  4 Hours: number analyzed (Participants) | 78 | 81 | 80 | 80
  4 Hours | -0.1 (2.13) | 2.6 (3.26) | 0.9 (3.14) | 1.1 (3.21)
  8 Hours: number analyzed (Participants) | 77 | 78 | 78 | 78
  8 Hours | 0.5 (2.10) | 2.5 (3.06) | 1.2 (2.78) | 0.7 (2.73)
  24 Hours: number analyzed (Participants) | 75 | 73 | 76 | 77
  24 Hours | 2.2 (2.59) | 4.0 (2.64) | 3.0 (2.72) | 3.2 (2.98)
  48 Hours: number analyzed (Participants) | 75 | 72 | 75 | 77
  48 Hours | 3.5 (2.60) | 4.9 (2.33) | 3.5 (3.00) | 4.1 (2.89)

3. Secondary Outcome: NRS Mean Pain Intensity Score at 4, 8, 24 and 48 Hours After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug administration) and at multiple time points up to 48 hours after Time 0 (time of administration of the first dose of study drug). A lower value indicates improvement in pain.
Time Frame: 4, 8, 24 and 48 hours after Time 0
Population: All randomized participants from the ITT Population with data available at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
units on a scale
  4 Hours: number analyzed (Participants) | 78 | 81 | 80 | 80
  4 Hours | 6.5 (2.45) | 4.1 (3.46) | 5.5 (3.24) | 5.6 (3.24)
  8 Hours: number analyzed (Participants) | 77 | 78 | 78 | 78
  8 Hours | 5.9 (2.51) | 4.2 (2.76) | 5.1 (2.75) | 5.9 (2.57)
  24 Hours: number analyzed (Participants) | 75 | 73 | 76 | 77
  24 Hours | 4.2 (2.67) | 2.7 (2.39) | 3.4 (2.55) | 3.4 (2.68)
  48 Hours: number analyzed (Participants) | 75 | 72 | 75 | 77
  48 Hours | 2.9 (2.60) | 1.9 (1.95) | 2.8 (2.65) | 2.6 (2.56)

4. Secondary Outcome: NRS SPID Over 4 Hours (SPID-4), 8 Hours (SPID-8) and 24 Hours (SPID-24) After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points up to 48 hours after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [max=10 at each time point] and negative numbers indicate an increase in pain [min=-10 at each time point]. The overall min and max are -10 and 10 times the number of hours specified: SPID-4=(-40 to 40), SPID-8=(-80 to 80) and SPID-24=(-240 to 240). The NRS SPID-4, 8 and 24 were analyzed using an ANCOVA model which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Baseline and 0 to 4, 0 to 8 and 0 to 24 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) Population who did not have missing SPID values.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 78 | 81 | 80 | 82
units on a scale
  SPID-4: number analyzed (Participants) | 78 | 81 | 80 | 80
  SPID-4 | 0.67 (1.036) | 7.70 (1.013) | 3.67 (1.023) | 3.74 (1.020)
  SPID-8: number analyzed (Participants) | 77 | 78 | 78 | 78
  SPID-8 | 1.32 (1.851) | 17.57 (1.835) | 8.26 (1.843) | 7.08 (1.837)
  SPID-24: number analyzed (Participants) | 75 | 73 | 76 | 77
  SPID-24 | 24.16 (5.001) | 75.67 (5.066) | 48.85 (4.962) | 44.17 (4.920)

5. Secondary Outcome: Total Pain Relief (TOTPAR) Over 4, 8, 24 and 48 Hours After Time 0
Description: TOTPAR was assessed by the participant using a 5-point NRS (0=no relief, 1=a little, 2=some, 3=a lot, 4=complete relief). TOTPAR scores were collected at Baseline (prior to study drug) and at multiple time points up to 48 hours after Time 0 (first dose of study drug). The TOTPAR scores are the sum of the pain relief at each time point multiplied by the duration in hours since the previous time point. Larger positive numbers indicate more pain relief (maximum=4 at each time point) and smaller positive numbers indicate less pain relief (minimum=0 at each time point). The overall minimum is 0 for each variable and the overall maximum is 4 times the number of hours specified for the variable: TOTPAR-4=(0 to 16), TOTPAR-8=(0 to 32), TOTPAR-24=(0 to 96) and TOTPAR-48=(0 to 192). TOTPAR-4, TOTPAR-8, TOTPAR-24 and TOTPAR-48 were analyzed using an ANCOVA model with factors for treatment, site and baseline pain intensity.
Time Frame: 4, 8, 24 and 48 hours after Time 0
Population: All randomized participants from the ITT Population with data available at each timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
units on a scale
  TOTPAR-4: number analyzed (Participants) | 78 | 81 | 80 | 80
  TOTPAR-4 | 2.50 (0.467) | 6.23 (0.457) | 4.07 (0.461) | 4.38 (0.460)
  TOTPAR-8: number analyzed (Participants) | 77 | 78 | 78 | 78
  TOTPAR-8 | 5.48 (0.848) | 13.85 (0.841) | 9.22 (0.845) | 8.95 (0.842)
  TOTPAR-24: number analyzed (Participants) | 75 | 73 | 76 | 77
  TOTPAR-24 | 27.33 (2.304) | 53.30 (2.334) | 40.50 (2.286) | 40.45 (2.267)
  TOTPAR-48: number analyzed (Participants) | 75 | 72 | 75 | 77
  TOTPAR-48 | 73.88 (4.684) | 118.12 (4.780) | 95.73 (4.680) | 100.15 (4.607)

6. Secondary Outcome: Time to Onset of Analgesia
Description: Time to onset of analgesia was measured as time to first perceptible pain relief confirmed by meaningful pain relief using the 2-stopwatch method. The study staff started 2 stopwatches as soon as the first dose of study drug was administered. Each participant was instructed to stop the first stopwatch when he or she experienced any perceptible pain relief and the second stopwatch when he or she experienced pain relief that was meaningful to them. If the second stopwatch was not stopped, time was censored at the time of the second dose of study drug or the use of rescue medication, whichever came first. If both stopwatches were not stopped time was censored at the time of the second dose of study drug or the use of rescue medication whichever came first. Time to onset of analgesia was defined as the time when the first stopwatch was stopped given that the second stopwatch is stopped.
Time Frame: From Time 0 (first dose of study drug) to time of confirmed meaningful pain relief (up to 64 minutes)
Population: All randomized participants from the ITT Population.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
minutes | NA [NA to NA] — Not estimable because less than 50% of participants achieved onset | 43.0 [21.0 to 64.0] | NA [43.0 to NA] — Not estimable because less than 50% of participants achieved onset | NA [41.0 to NA] — Not estimable because less than 50% of participants achieved onset

7. Secondary Outcome: Percentage of Participants With Scores in Each Pain Relief Category at 4, 8, 24 and 48 Hours After Time 0
Description: Pain relief was assessed by the participant using a 5-point NRS (0=no relief, 1=a little, 2=some, 3=a lot, 4=complete relief). The percentage of participants with scores in each pain relief category are reported. Missing values were imputed.
Time Frame: 4, 8, 24 and 48 hours after Time 0 (first dose of study drug)
Population: All randomized participants from the ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
percentage of participants
  4 Hours - No relief | 60.8 | 24.7 | 43.8 | 41.5
  4 Hours - A little relief | 21.5 | 16.0 | 22.5 | 23.2
  4 Hours - Some relief | 13.9 | 21.0 | 13.8 | 11.0
  4 Hours - A lot of relief | 1.3 | 19.8 | 13.8 | 13.4
  4 Hours - Complete relief | 1.3 | 18.5 | 6.3 | 8.5
  8 Hours - No relief | 43.0 | 18.5 | 32.5 | 32.9
  8 Hours - A little relief | 35.4 | 14.8 | 22.5 | 28.0
  8 Hours - Some relief | 7.6 | 27.2 | 21.3 | 18.3
  8 Hours - A lot of relief | 10.1 | 23.5 | 12.5 | 12.2
  8 Hours - Complete relief | 1.3 | 12.3 | 8.8 | 3.7
  24 Hours - No relief | 20.3 | 6.2 | 7.5 | 11.0
  24 Hours - A little relief | 19.0 | 2.5 | 21.3 | 12.2
  24 Hours - Some relief | 29.1 | 23.5 | 25.0 | 19.5
  24 Hours - A lot of relief | 17.7 | 38.3 | 26.3 | 39.0
  24 Hours - Complete relief | 8.9 | 19.8 | 15.0 | 12.2
  48 Hours - No relief | 17.7 | 2.5 | 8.8 | 4.9
  48 Hours - A little relief | 13.9 | 8.6 | 11.3 | 6.1
  48 Hours - Some relief | 20.3 | 12.3 | 20.0 | 20.7
  48 Hours - A lot of relief | 27.8 | 38.3 | 32.5 | 35.4
  48 Hours - Complete relief | 15.2 | 27.2 | 21.3 | 26.8

8. Secondary Outcome: Percentage of Participants With Peak Scores in Each Pain Relief Category
Description: Peak pain relief is the highest value of pain relief experienced during the study. Pain relief was assessed by the participant using a 5-point NRS (0=no relief, 1=a little, 2=some, 3=a lot, 4=complete relief). The percentage of participants with peak scores in each pain relief category are reported.
Time Frame: From Time 0 (first dose of study drug) up to 48 hours
Population: All randomized participants from the ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
percentage of participants
  No relief | 6.3 | 0 | 1.3 | 3.7
  A little relief | 11.4 | 2.5 | 3.8 | 1.2
  Some relief | 19.0 | 9.9 | 12.5 | 13.4
  A lot of relief | 36.7 | 42.0 | 46.3 | 40.2
  Complete relief | 26.6 | 45.7 | 36.3 | 41.5
  A lot of relief + Complete relief | 63.3 | 87.7 | 82.6 | 81.7

9. Secondary Outcome: Time to Peak Pain Relief
Description: Time to peak pain relief is the time to the highest value of pain relief experienced during the study. Pain relief was assessed by the participant using a 5-point NRS (0=no relief, 1=a little, 2=some, 3=a lot, 4=complete relief). If no pain relief was observed, then the time was censored at the time of the last pain assessment.
Time Frame: From Time 0 (first dose of study drug) to time of peak pain relief (up to 1437 minutes)
Population: All randomized participants from the ITT Population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
minutes | 1200.0 [720.0 to 1200.0] | 360.0 [181.0 to 719.0] | 720.0 [420.0 to 960.0] | 1200.0 [720.0 to 1437.0]

10. Secondary Outcome: Time to First Perceptible Pain Relief
Description: Time to first perceptible pain relief was evaluated using the 2 stopwatch method and is defined as the time when the participant stops the first stopwatch. If it was not stopped time was censored at the time that the second stopwatch was stopped or the time of the second dose or the time that rescue medication was used whichever came first.
Time Frame: From Time 0 (first dose of study drug) to time of first perceptible pain relief (up to 83 minutes)
Population: All randomized participants from the ITT Population.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
minutes | 29.0 [6.0 to 83.0] | 23.0 [10.0 to 43.0] | 15.0 [11.0 to 42.0] | 27.0 [14.0 to 74.0]

11. Secondary Outcome: Time to Meaningful Pain Relief
Description: Time to meaningful pain relief was evaluated using the 2 stopwatch method and is defined as the time when the participant stops the second stopwatch. If it was not stopped time was censored at the time that the second stopwatch was stopped or the time of the second dose or the time that rescue medication was used whichever came first.
Time Frame: From Time 0 (first dose of study drug) to time of meaningful pain relief (up to 227 minutes)
Population: All randomized participants from the ITT Population.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
minutes | 238.0 [121.0 to NA] — Not estimable because less than 50% of participants achieved meaningful pain relief | 92.0 [79.0 to 120.0] | 122.0 [90.0 to 227.0] | 166.0 [87.0 to 240.0]

12. Secondary Outcome: Percentage of Participants Using Rescue Medication for Pain
Description: The percentage of participants who needed to take an alternate medication for pain relief during the treatment period.
Time Frame: From Time 0 (first dose of study drug) up to 48 hours
Population: All randomized participants from the ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
percentage of participants | 97.5 | 55.6 | 87.5 | 87.8

13. Secondary Outcome: Time to First Use of Rescue Medication for Pain
Description: Time to first use of rescue medication is the time from Time 0 (time of administration of the first dose of study drug) to the first use of rescue medication. If rescue medication was not taken the time was censored at the time of the last pain assessment.
Time Frame: From Time 0 to time of first use of rescue medication (up to 280 minutes)
Population: All randomized participants from the ITT Population.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
minutes | 107.0 [77.0 to 125.0] | 937.0 [349.0 to NA] — Not estimable because too few participants used rescue medication | 219.5 [105.0 to 260.0] | 193.0 [92.0 to 280.0]

14. Secondary Outcome: Total Use of Rescue Medication Over 0 to 24 Hours and 0 to 48 Hours
Description: Total use of rescue medication is defined as the number of times a participant took rescue medication.
Time Frame: Over 24 and 48 hours after Time 0 (first dose of study drug)
Population: All randomized participants from the ITT Population who used rescue medication during the specified time intervals.
Measure: Mean (Standard Deviation); unit: number of uses
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 77 | 45 | 70 | 72
number of uses
  0-24 Hours: number analyzed (Participants) | 77 | 41 | 68 | 71
  0-24 Hours | 3.8 (1.98) | 2.2 (1.69) | 2.6 (1.62) | 2.9 (1.67)
  0-48 Hours | 5.6 (3.60) | 2.9 (2.81) | 3.7 (2.68) | 3.9 (2.69)

15. Secondary Outcome: Participant's Global Evaluation of Study Drug
Description: Global evaluation of study drug was completed at the end of treatment (Day 3) or before early termination if a participant discontinued early. Participants were asked to provide an overall rating of their study medication in controlling pain on a 5-point NRS, where 0=poor, 1=fair, 2=good, 3=very good, and 4=excellent. The percentage of participants with scores in each pain relief category are reported.
Time Frame: End of treatment (Day 3) or early termination
Population: All randomized participants from the ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Number analyzed (Participants) | 79 | 81 | 80 | 82
percentage of participants
  Poor | 25.3 | 2.5 | 5.0 | 14.6
  Fair | 25.3 | 7.4 | 16.3 | 15.9
  Good | 19.0 | 16.0 | 26.3 | 14.6
  Very Good | 19.0 | 32.1 | 30.0 | 24.4
  Excellent | 10.1 | 38.3 | 18.8 | 28.0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to the Follow-up visit (up to 9 days).
Arm/Group | Placebo | Buprenorphine 0.5 mg TID | Buprenorphine 0.25 mg TID | Buprenorphine 0.125 mg TID
Serious Adverse Events (participants affected / at risk) | 0/79 | 1/81 | 0/80 | 0/82
Other Adverse Events (participants affected / at risk) | 38/79 | 76/81 | 67/80 | 57/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Buprenorphine 0.5 mg TID (N=81) | Buprenorphine 0.25 mg TID (N=80) | Buprenorphine 0.125 mg TID (N=82)
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Buprenorphine 0.5 mg TID (N=81) | Buprenorphine 0.25 mg TID (N=80) | Buprenorphine 0.125 mg TID (N=82)
Nausea (Gastrointestinal disorders) | 13 | 68 | 47 | 36
Vomiting (Gastrointestinal disorders) | 4 | 59 | 33 | 24
Constipation (Gastrointestinal disorders) | 1 | 8 | 6 | 9
Dizziness (Nervous system disorders) | 7 | 44 | 26 | 18
Headache (Nervous system disorders) | 9 | 13 | 23 | 15
Somnolence (Nervous system disorders) | 0 | 11 | 6 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 11 | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 8 | 1 | 2
Oxygen saturation decreased (Investigations) | 4 | 7 | 8 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 7 | 0 | 0
Hot flush (Vascular disorders) | 1 | 5 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No